CLINICAL TRIAL: NCT07113652
Title: Exploring the Efficacy of Temporal Interference Stimulation in the Treatment of Obsessive-Compulsive Disorder
Brief Title: The Efficacy of Temporal Interference Stimulation in the Treatment of Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-018
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nucleus Accumbens Group(NAcc)-Bed Nucleus of the Stria Terminalis Group(BNST)-Exploratory group (Other): Participants assigned to NAcc-BNST group will receive stimulation targeting the NAcc in Phase 1 and the BNST in Phase 2. During the exploratory phase, based on participants' preferences, they will be randomly allocated to receive stimulation targeting one of the following regions: the caudate nucleus, the putamen, or the amygdala.
  Interventions: Device: TI stimulation device (nerviox-1000）
- Bed Nucleus of the Stria Terminalis Group(BNST)-Nucleus Accumbens Group(NAcc)-Exploratory group (Other): Participants assigned to BNST-NAcc group will receive stimulation targeting the BNST in Phase 1 and the NAcc in Phase 2. During the exploratory phase, based on participants' preferences, they will be randomly allocated to receive stimulation targeting one of the following regions: the caudate nucleus, the putamen, or the amygdala.
  Interventions: Device: TI stimulation device (nerviox-1000）
- Sham Group-NAcc Group or BNST Group-Exploratory group (Other): Participants assigned to the Sham-NAcc or Sham-BNST groups will receive sham stimulation in Phase 1, followed by active stimulation targeting the NAcc or the BNST in Phase 2. During the exploratory phase, based on participants' preferences, they will be randomly allocated to receive stimulation targeting one of the following regions: the caudate nucleus, the putamen, or the amygdala.
  Interventions: Device: TI stimulation device (nerviox-1000）

INTERVENTIONS:
Device: TI stimulation device (nerviox-1000） — The TI stimulation device (nerviox-1000) delivers temporally interfering electrical fields with a 130 Hz envelope frequency, generated by high-frequency carrier waves. The stimulation is applied for 20 minutes per session, with a peak current of 3-4 mA per channel, adjusted based on individual tolerance. The stimulation targets include the nucleus accumbens, bed nucleus of the stria terminalis, amygdala, caudate nucleus, and putamen. Stimulation is administered twice daily, with each treatment phase lasting 7 consecutive days.
  Sham stimulation uses identical electrode placement and setup as active stimulation. A brief 30-second ramp-up is applied to mimic real stimulation, followed by rapid reduction to 0 mA or minimal current. A 1 mA "tail" current is delivered in the final 30 seconds to simulate the tapering effect of active stimulation.

SUMMARY:
This study aims to evaluate the efficacy of Temporal Interference (TI) stimulation in treating patients with obsessive-compulsive disorder (OCD) and to explore its potential neural mechanisms using magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
This randomized, blind, multi-phase clinical trial aims to evaluate the efficacy of Temporal Interference (TI) stimulation in patients with treatment obsessive-compulsive disorder (OCD), and to compare the effects of stimulating different brain regions.

The study includes three phases:

* Phase 1: Patients are randomly assigned to receive either sham stimulation, bilateral nucleus accumbens (NAcc) stimulation, or bilateral bed nucleus of the stria terminalis (BNST) stimulation.
* Phase 2: Non-responders from Phase 1 enter a second phase, receiving stimulation to the opposite target region. Sham participants are re-randomized to NAcc or BNST.
* Phase 3 (Exploratory): Remaining non-responders may opt to receive stimulation targeting the caudate nucleus, the putamen, or the amygdala.

Stimulation is delivered twice daily for 7 days in each phase, followed by follow-up assessments for up to 4 weeks. Comprehensive clinical assessments, self-reported symptom scales, magnetic resonance imaging (MRI), electroencephalography (EEG), and cognitive function tests are conducted before and after each phase to ensure data consistency. Additionally, clinical assessments and self-reported scales are repeated 1 week after the end of each treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Diagnosis of OCD per DSM-5
* Y-BOCS score ≥20
* Have a documented history of at least two adequate trials of selective serotonin reuptake inhibitors (SSRIs). If currently receiving SSRI treatment, the dosage must be stable for at least 8 weeks prior to enrollment
* With at least 9 years of education

Exclusion Criteria:

* Any DSM-5 diagnosis other than OCD (except OCPD)
* OCD symptoms too severe to complete assessments
* Received electroconvulsive therapy (ECT) within the past 6 months
* Received other forms of neuromodulation within the past 2 months（see Item 3 for ECT）
* Severe medical illness or seizure risk (e.g., cardiovascular, respiratory conditions)
* Neurological disorders or history of brain injury/surgery
* MRI-incompatible implants (e.g., pacemaker, stents, cochlear implants).
* Current suicidal risk per investigator judgment
* Pregnant or planning pregnancy during the study
* Started structured OCD psychotherapy within 3 months, with expected change during treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms improvement | phase-specific baseline and 1 week after the end of each phase of TI treatment
  The severity of OCD symptoms is assessed using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). Obsessive-compulsive symptoms improvement is reflected by Y-BOCS reduction rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China